CLINICAL TRIAL: NCT03324594
Title: A Pilot Functional Performances Study of The Wondaleaf-Cap and The Wondaleaf-On-Man Synthetic Male Condom
Brief Title: A Pilot Functional Performances Study of Two Synthetic Male Condom
Acronym: WONDALEAF-MEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Twin Catalyst Sdn. Bhd. (Industry); Sarawak Research Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: NMRR-17-1895-37590
Record Dates: First submitted 2017-09-24; First posted 2017-10-27 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Functional Performance; Synthetic Male Condom
Keywords: functional performance; synthetic male condom

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Throughout the study, neither participating couples, clinic staff, research assistants or researchers are masked to condom assignment as there are observable differences on packaging and design between the test condom (WLC and WLM) and the control condom (durex-Together). However, statisticians, sponsors, and medical reviewers are masked until completion of the final report to minimize biases potentially emerge during data analyses and results reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Active Comparator): Participants will be first given (1) WONDALEAF-CAP, followed by (2) WONDALEAF-ON-MEN, and last with (3) durex-TOGETHER after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)
- Group B (Active Comparator): Participants will be first given (1) WONDALEAF-CAP, followed by (2) durex-TOGETHER, and last with (3) WONDALEAF-ON-MEN after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)
- Group C (Active Comparator): Participants will be first given (1) WONDALEAF-ON-MEN, followed by (2) durex-TOGETHER, and last with (3) WONDALEAF-CAP after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)
- Group D (Active Comparator): Participants will be first given (1) WONDALEAF-ON-MEN, followed by (2) WONDALEAF-CAP, and last with (3) durex-TOGETHER after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)
- Group E (Active Comparator): Participants will be first given (1) durex-TOGETHER, followed by (2) WONDALEAF-ON-MEN, and last with (3) WONDALEAF-CAP after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)
- Group F (Active Comparator): Participants will be first given (1) durex-TOGETHER, followed by (2) WONDALEAF-CAP, and last with (3) WONDALEAF-ON-MEN after completion of four times usage for each condom type. The participants will be asked to complete four times of usage for each condom type within three to four months. There will be a baseline survey before the use of the first condom type, and subsequent evaluations upon completion of each condom type.
  Interventions: Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator)

INTERVENTIONS:
Device: (1) WONDALEAF-CAP, (2) WONDALEAF-ON-MEN, (3) durex-TOGETHER (active comparator) — 1. WONDALEAF-ON-MEN (WLM) is a polyurethane pouch with outstretching adhesive shield. The pouch covers the penis in man user; while the adhesive shield covers the groin regions to provide extra protection for the couples. The pouch is equivalent to marketed polyurethane male; while the adhesive shield is equivalent to marketed polyurethane wound dressing. WLM integrally joined with an adhesive wound dressing, both made of the same polyurethane material.
  2. WONDALEAF-CAP (WLC) is a miniature form of WLM: the pouch covers glans penis and the adhesive shield wraps around the shaft of the penis only, thereby emulating the configuration of a donned regular condom on the penis. Because of the adhesive coating, WLC overcomes the problems of slippage when the penis is flaccid.
  3. The durex-TOGETHER serves as the active comparator in this study. It is a transparent natural rubber latex male condom which is commercially available.

SUMMARY:
Over the decades, male condoms had been widely commercialized and used to protect against unintended pregnancy and sexually transmitted infections (STI). While natural rubber latex (NRL) male condoms has majority proportion of male condoms in the market, synthetic male condoms (SMC) made from polyurethane or other synthetic materials remain new to the consumers. Notably, synthetic male condoms are found to be more durable, non-allergenic and have better compatibility with lubricants when compared to NRL male condoms. The SMCs that have FDA approval and commercially available are AvantiTM (polyisoprene condom), Trojan SupraTM (polyurethane condom) and eZ.onTM (polyurethane condom). Although the effectiveness of SMCs in the prevention of sexually transmitted infections has yet to be established, SMCs are believed to be comparable to NRL male condoms in both STI prevention and contraception protection. Notwithstanding, a recent literature had reported the shortfall on the quality of variant male condoms in the market, especially nonconforming volumetric capacity, burst pressure and freedom from holes. This warrant the current investigation, to evaluate the functional performances of two newly invented synthetic male condoms, branded as "WONDALEAF-CAP" (WLC) and "WONDALEAF-ON-MAN" (WLM). Apart from being made of polyurethane, the major feature of WLC and WLM are nonetheless their adhesive coating on the outer rim of the condom opening which by securely adhering to the foreskin, prevent slippage of condom and spillage of male ejaculate or secretions when the penis is flaccid, and thereby improve the user-friendliness of condom usage.

ELIGIBILITY:
Inclusion Criteria:

1. Their female sexual partners are not at risk of pregnancy (using alternate contraception);
2. They don't have known sexually transmitted infections, including HIV/AIDS;
3. They should be experienced condom users, minimum 10 male condoms used in the last 12 months;
4. They are between 18 to 45 years of age;
5. They are in a monogamous heterosexual relationship and agree to practice vaginal sex only using male condoms provided by the study.

Exclusion Criteria:

1. couples who work for the research team or who are close relatives of the research team;
2. men with known allergy to natural rubber latex;
3. men with known sensitivity to the residual chemicals used in the manufacture of natural rubber latex condoms or the test condom materials;
4. couples where one knowingly has a sexually transmitted infection.
5. couples who are pregnant in time of recruitment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to the nature of the studied intervention (male condom), only male respondents who fulfill the inclusion and exclusion criteria will be eligible for participation.
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical Slippage Rates (CSR) | Through study completion, an average of 3 months. In specific, CSR will be evaluated within 24 hours after use of individual condom, for each condom type
  Number of condoms that slipped completely off the penis during intercourse or withdrawal, divided by the number of condoms used during intercourse; reported as a percentage.
Clinical Breakage Rates (CBR) | Through study completion, an average of 3 months. In specific, CBR will be evaluated within 24 hours after use of individual condom, for each condom type
  Number of condoms that broke during intercourse or withdrawal, divided by the number of condoms used during intercourse; reported as a percentage.
Clinical Failure Rates (CFR) | Through study completion, an average of 3 months. In specific, CFR will be calculated after completion of four times usage, for each condom type
  CFR is the sum of CSR and CBR for each condom type

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 3 months. In specific, it will be measured after completion of four times usage, for each condom type
  This outcome will reflect the safety of the male condoms used. Proportion of participants with symptoms of and proportion of condom uses with reports of individual complaints (eg. irritation, burning, itching, bleeding, etc.) during or immediately after any of the 3 separate uses will be calculated for each condom type. Adverse events will be classified by relatedness, expectedness and severity.
Comfort in use | Through study completion, an average of 3 months. In specific, it will be measured after completion of four times usage, for each condom type
  This will reflect the acceptability of the male condoms used. It is a self-reported comfortability on each type of male condoms used
Ease of insertion and removal | Through study completion, an average of 3 months. In specific, it will be measured after completion of four times usage, for each condom type
  This will reflect the acceptability of the male condoms used. It is a self-reported ease of insertion and removal for each type of male condoms used
Favorability of product attributes | Through study completion, an average of 3 months. In specific, it will be measured after completion of four times usage, for each condom type
  This will reflect the acceptability of the male condoms used. It is a self-reported favorability towards attributes of each male condoms' type used
Adequacy and feel of lubrication | Through study completion, an average of 3 months. In specific, it will be measured after completion of four times usage, for each condom type
  This will reflect the acceptability of the male condoms used. It is a self-reported adequacy and feel of lubrication for each type of male condoms used.

CONTACTS AND LOCATIONS:
Overall Officials: Chuo Yew Ting, BPharm., MPhil., Principal Investigator — (1) Sarawak Research Society, (2) Sarawak State Health Department, Ministry of Health
Locations (2):
- Malaysia (2):
  - Sarawak Family Planning Association, Kuching, Sarawak
  - Sarawak Research Society, Kuching, Sarawak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bounds W, Molloy S, Guillebaud J. Pilot study of short-term acceptability and breakage and slippage rates for the loose-fitting polyurethane male condom eZ.on bi-directional: a randomized cross-over trial. Eur J Contracept Reprod Health Care. 2002 Jun;7(2):71-8. PMID 12201325
- [Background] Duarte JT, de Almeida AE, de Mello Pereira Abrantes S. Quality evaluation of commercially available male condoms in Rio de Janeiro, Brazil, 2009-2011. Reprod Health. 2016 Dec 7;13(1):145. doi: 10.1186/s12978-016-0254-5. PMID 27923380
- [Background] Fontanet AL, Saba J, Chandelying V, Sakondhavat C, Bhiraleus P, Rugpao S, Chongsomchai C, Kiriwat O, Tovanabutra S, Dally L, Lange JM, Rojanapithayakorn W. Protection against sexually transmitted diseases by granting sex workers in Thailand the choice of using the male or female condom: results from a randomized controlled trial. AIDS. 1998 Oct 1;12(14):1851-9. doi: 10.1097/00002030-199814000-00017. PMID 9792386
- [Background] French PP, Latka M, Gollub EL, Rogers C, Hoover DR, Stein ZA. Use-effectiveness of the female versus male condom in preventing sexually transmitted disease in women. Sex Transm Dis. 2003 May;30(5):433-9. doi: 10.1097/00007435-200305000-00010. PMID 12916135
- [Background] Gallo MF, Grimes DA, Lopez LM, Schulz KF. Non-latex versus latex male condoms for contraception. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD003550. doi: 10.1002/14651858.CD003550.pub2. PMID 16437459
- [Derived] Ting CY, Ting RS, Lim CJ, King TL, Ting H, Gerofi J. Pilot study on functional performance and acceptability of two new synthetic adhesive male condoms (Wondaleaf): a randomized cross-over trial. Contraception. 2019 Jul;100(1):65-71. doi: 10.1016/j.contraception.2019.02.013. Epub 2019 Mar 11. PMID 30871936
- See also: ISO/WD 29943-1. Condoms - Guidance on clinical studies - Part 1: Male condoms, clinical function studies based on self-reports — http://www.iso.org/standard/62497.html